CLINICAL TRIAL: NCT06315634
Title: Prospective Randomized Controlled Clinical Trial to Compare Intrathecal Dexmedetomidine Versus Midazolame in Orthopedic Cancer Surgeries
Brief Title: Intrathecal Dexmedetomidine vs Midazolame
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Mohammed Said Nasef Zedan, assistant lecturer, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AP210330102
Record Dates: First submitted 2024-02-09; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Midazolam; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Heavy Bupivacaine plus normal saline (Active Comparator): 2.5 ml of 0.5% hyperbaric Bupivacaine plus 0.5 ml 0.9 % saline
  Interventions: Drug: Bupivacain
- Heavy Bupivacaine plus dexmedetomidine (Experimental): 2.5 ml of 0.5% hyperbaric Bupivacaine plus 5 micrograms dexmedetomidine in 0.5 ml 0.9 % saline
  Interventions: Drug: Dexmedetomidine; Drug: Bupivacain
- Heavy Bupivacaine plus midazolam (Experimental): 2.5 ml of 0.5% hyperbaric Bupivacaine plus 2 milligrams midazolam in 0.5 ml 0.9 % saline
  Interventions: Drug: Midazolam; Drug: Bupivacain

INTERVENTIONS:
Drug: Dexmedetomidine — 5 micrograms intrathecal dexmedetomidine
  Other Names: Spinal dexmedetomidine
  Arms: Heavy Bupivacaine plus dexmedetomidine
Drug: Midazolam — 2 milligrams intrathecal midazolam
  Other Names: Spinal midazolam
  Arms: Heavy Bupivacaine plus midazolam
Drug: Bupivacain — 12.5 milligrams 0.5% intrathecal hyperbaric bupivacaine
  Other Names: Spinal bupivacaine

SUMMARY:
Prospective Randomized Controlled Clinical Trial to Compare Intrathecal Dexmedetomidine Versus Midazolame in Orthopedic Cancer Surgeries

DETAILED DESCRIPTION:
Comparison of intrathecal dexmedetomidine plus Bupivacaine vs intrathecal midazolam plus Bupivacaine on duration of sensory and motor blockade and hemodynamic parameters of patients

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lower limb orthopedic cancer surgery.
* ASA I, II, III.
* Age 20 to 70 year
* Healthy volunteers

Exclusion Criteria:

* Age less than 20 and older than 70.
* ASA IV, V.
* patients' refusal.
* patients with coagulopathy.
* patients with severe valvular stenosis
* patients with infection at site of injection

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Duration of sensory block | 12 hours
  Duration of sensory block after spinal anesthesia by the ability of the patient to demonstrate the pinprick sensation

SECONDARY OUTCOMES:
Incidence of vomiting occurrence | 12 hours
  The patient will be reported in case of vomiting occurrence
Sedation | 12 hours
  Ramsay's sedation score1: anxious, agitated and restlessness, 2: oriented and cooperative, 3: responds to command only, 4: brisk response to loud voice and light glabellar tap, 5: sluggish to no response to light glabellar tap or loud auditory stimulus, 6: no response even to pain
Change in mean arterial blood pressure | 12 hours
  Non invasive blood pressure measurement
Duration of motor block | 12 hours
  Ability of patient to regain full motor power
Change in heart rate | 12 hours
  Heart rate will be compared between the three groups and will be compared with baseline preoperative values in each group

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Elwasef, MD, Study Director — NCI Egypt
Locations (1):
- National cancer institute, Cairo, Egypt